CLINICAL TRIAL: NCT00231543
Title: Laparoscopy in Children: Does it Decrease the Metabolic, Endocrine and Inflammatory Stress Response to Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99SG92
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2005-10

CONDITIONS: Gastro-Oesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

INTERVENTIONS:
Procedure: Laparoscopic fundoplication
Procedure: open Nissen fundoplication

SUMMARY:
The aim of this trial was to characterise the intra and post operative metabolic, endocrine and inflammatory response to laparoscopic fundoplication in children. We are testing the hypothesis that laparoscopic fundoplication is associated with a lack of hypermetabolism and catabolism and blunting of the endocrine/inflammatory stress response

ELIGIBILITY:
Inclusion Criteria:

* infants and children with gastro-oesophageal reflux

Exclusion Criteria:

* septic shock, multi-organ dysfunction syndrome, cardiac, renal or congenital metabolic abnormalities

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

PRIMARY OUTCOMES:
resting energy expenditure

SECONDARY OUTCOMES:
whole body protein turnover
indices of inflammatory response
pro and anti inflammatory cytokines
free radical production
post operative pain

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Pierro, Prof, Principal Investigator — Institute of Child Health
Locations (1):
- Great Ormond Street Hospital and the Institute of Child health, London, United Kingdom

REFERENCES:
- [Derived] McHoney M, Wade AM, Eaton S, Howard RF, Kiely EM, Drake DP, Curry JI, Pierro A. Clinical outcome of a randomized controlled blinded trial of open versus laparoscopic Nissen fundoplication in infants and children. Ann Surg. 2011 Aug;254(2):209-16. doi: 10.1097/SLA.0b013e318226727f. PMID 21725231
- [Derived] McHoney M, Eaton S, Wade A, Carnielli V, Kiely E, Drake D, Curry J, Pierro A. Effect of laparoscopy and laparotomy on energy and protein metabolism in children: a randomized controlled trial. J Pediatr. 2010 Sep;157(3):439-44, 444.e2. doi: 10.1016/j.jpeds.2010.02.067. Epub 2010 Apr 18. PMID 20400097